CLINICAL TRIAL: NCT07052071
Title: Impact of Transcatheter Aortic Valve Implantation (TAVI) on the Gut Microbiota in Patients With Aortic Valve Stenosis
Acronym: GUT-TAVI
Status: Recruiting | Type: Observational
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, Professor of Cardiology, Hippocration General Hospital
Other Study IDs: GUT-TAVI
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Aortic Stenosis; Gut Microbiome; Gut Microbiota; TAVI; TAVI(Transcatheter Aortic Valve Implantation)
Keywords: TAVI
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (TMAO and other biochemical markers) without DNA analysis. Stool with DNA extraction for 16S rRNA sequencing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVI
  Interventions: Procedure: TAVI

INTERVENTIONS:
Procedure: TAVI — Transcatheter Aortic Valve Implantation (TAVI) is a minimally invasive method for replacing the aortic valve in patients with severe aortic stenosis. The procedure involves the placement of a bioprosthetic valve within the patient's degenerated aortic valve via a catheter.

SUMMARY:
This study investigates the impact of transcatheter aortic valve implantation (TAVI) on the composition and function of the gut microbiota in patients with severe aortic valve stenosis. The improvement in haemodynamics following TAVI may positively influence gut microbial balance by increasing splanchnic perfusion and reducing intestinal congestion. A total of 40 patients undergoing TAVI at the "Hippokration" General Hospital of Athens will be enrolled, with the aim of analysing stool and blood samples before and after the procedure. The primary endpoint is the change in gut microbiota composition two months post-TAVI, assessed via 16S rRNA sequencing. Secondary endpoints include changes in serum TMAO levels and their association with the severity of aortic stenosis and post-procedural valve haemodynamics. Data will be collected at two timepoints (1 month up to 1 day pre-TAVI and 3 to 4 months post-TAVI), along with dietary questionnaires to account for potential confounding factors. This observational study aims to highlight the potential relationship between cardiac function and the gut microbiome, offering new perspectives for targeted therapeutic strategies in cardiovascular disease.

DETAILED DESCRIPTION:
Hypothesis The interaction between transcatheter aortic valve implantation (TAVI) and the gut microbiota represents an emerging field of investigation with potential clinical implications. Beyond restoring haemodynamic function, TAVI may influence the composition and function of the gut microbiome through several mechanisms. Improved cardiac output following TAVI enhances splanchnic perfusion, potentially reducing mucosal oedema and congestion, which may restore intestinal permeability and lead to favourable changes in microbiome composition.

Study Objective To evaluate changes in the gut microbiota following TAVI in patients with severe aortic valve stenosis.

Study Timeline and Data Collection Phase 1: Screening and Baseline Data Collection (1 month to 24 hours before TAVI, T1) Participants will be assessed for eligibility based on inclusion/exclusion criteria. Informed consent will be obtained, and participants will agree to telephone follow-up.

Collected data will include:

* Demographics and anthropometrics: sex, age, weight, height, BMI
* Social history: smoking, alcohol, substance use
* Medical history: comorbidities including hypertension, diabetes, dyslipidaemia, vascular disease, heart failure, stroke, TIA, embolism, PE
* Echocardiography parameters
* Venous Blood Sample (T1):

Collected up to 24 hours before TAVI for the following markers: TMAO, Complete blood count, Liver enzymes (SGOT, SGPT, ALP, γ-GT), Renal function (urea, creatinine), Electrolytes (K⁺, Na⁺, Ca²⁺, Mg²⁺), NT-proBNP, hsCRP, eGFR using the Cockcroft-Gault equation.

- Stool Sample & Dietary Assessment (T1): Participants will collect a stool sample using a standardised kit for 16S rRNA sequencing. A food frequency questionnaire will be completed to account for dietary influences on microbiota. This questionnaire will be repeated at each sample collection.

Sample Collection Procedure:

Participants will follow hygiene protocols and use provided containers for stool collection. Samples will be labeled with study ID, sample sequence (A or B), date of collection, and procedure type, and will be returned to the hospital promptly. No identifiable information will be recorded on the specimen.

Phase 2: Follow-Up (3-4 months after TAVI, T2) All assessments will be repeated 3 months post-procedure. If antibiotics were taken within this period, the follow-up assessment will be delayed by 1 month (i.e., 4 months post-TAVI).

Timepoint Comparisons:

T1 vs T2: Assess the impact of TAVI on gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Aortic stenosis suitable for TAVI

Exclusion Criteria:

Patients will be excluded if they present any condition or intervention that may independently affect gut microbiota composition. These include:

* Use of antibiotics, systemic corticosteroids, antivirals, probiotics, bile acid sequestrants, or new medications within one month prior to enrollment.
* History of inflammatory bowel disease.
* End-stage renal disease requiring dialysis.
* End-stage chronic liver disease.
* Acute infection. Patients with aortic stenosis due to rheumatic fever or infectious endocarditis will be excluded.
* Active cancer under treatment.
* Psychiatric illness impairing ability to consent.
* Substance or alcohol abuse.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include 40 patients undergoing clinically indicated TAVI at the Hemodynamic Laboratory of the "Hippokration" General Hospital of Athens. This sample size is considered sufficient based on the limited available literature. Interim analysis will be conducted after the first 10 patients have completed the study to reassess and, if necessary, adjust the final sample size. Written informed consent is a prerequisite for inclusion.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiota composition (via 16S rRNA sequencing) | 3 months post TAVI

SECONDARY OUTCOMES:
Change in serum trimethylamine N-oxide (TMAO) levels | 3 months post TAVI
Correlation of microbiota changes with severity of aortic stenosis at baseline | 3 months post TAVI
Correlation of microbiota changes with haemodynamic parameters | 3 months post TAVI

CONTACTS AND LOCATIONS:
Locations (1):
- Hippokration General Hospital of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided